CLINICAL TRIAL: NCT01539941
Title: Family-Based Protocol for Medication Integration in Treatment of Comorbid ASU/ADHD in Routine Care
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The National Center on Addiction and Substance Abuse at Columbia University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: R21DA031305-01A1 (NIH)
Record Dates: First submitted 2012-02-15; First posted 2012-02-28 (Estimated); Last update posted 2015-08-04 (Estimated); Status verified 2012-02

CONDITIONS: Adolescent Substance Abuse; Attention Deficit Hyperactivity Disorder
Keywords: Co-occurring adolescent substance use and ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Medication Integration Protocol (Experimental)
  Interventions: Behavioral: Medication integration protocol

INTERVENTIONS:
Behavioral: Medication integration protocol — MIP is a 5 session protocol. The first session consists of pretreatment assessment activities using measures administered during routine clinical intake. The following sessions, MIP Sessions 1-4, are meant to be delivered sequentially, commencing sometime after session 2 or 3 of treatment, that is, after completion of initial treatment contracting and engagement interventions that will usually be focused on ASU-related referral problems for this population. The proposed pilot work will shed light on the optimal timing for MIP Sessions 1-4.

SUMMARY:
The goal of this proposal is to develop and pilot a brief protocol designed to systematically integrate pharmacological interventions for attention deficit hyperactivity disorder (ADHD) into behavioral treatment services for adolescent substance users with comorbid ADHD in everyday care. ADHD is a prevalent co-occurring condition for adolescent substance use (ASU) that can significantly impede successful ASU treatment but is vastly under-diagnosed and undertreated among ASU clients in agency settings. Moreover, ADHD medication acceptance and compliance is particularly difficult to achieve in high-risk adolescent populations.

DETAILED DESCRIPTION:
The goal of this proposal is to develop and pilot a brief protocol designed to systematically integrate pharmacological interventions for attention deficit hyperactivity disorder (ADHD) into behavioral treatment services for adolescent substance users with comorbid ADHD in everyday care. ADHD is a prevalent co-occurring condition for adolescent substance use (ASU) that can significantly impede successful ASU treatment but is vastly under-diagnosed and undertreated among ASU clients in agency settings. Moreover, ADHD medication acceptance and compliance is particularly difficult to achieve in high-risk adolescent populations. The proposed R21 study will use an interrupted time series design to test a brief protocol designed to promote integration of evidence-based ADHD pharmacotherapy into routine behavioral services for ASU: Medication Integration Protocol (MIP). MIP is a 5-session family-based protocol delivered during the early portion of ASU treatment that contains three research-based elements: (1) standardized psychiatric assessment and family-focused psychoeducation about adolescent ADHD; (2) an approved ADHD medication regimen (OROS-MPH) with demonstrated efficacy for ASU/ADHD clients; (3) family-based interventions to support medication acceptance (as indicated) and coordination of care between psychiatric and behavioral services. MIP will be integrated into existing family-based services at one partnering clinical site: 20 ASU/ADHD cases will be treated by site family therapists who will be newly trained and monitored in MIP. The partnering clinic provides family therapy as the routine standard of care for outpatient behavioral health and offers on-site child psychiatry services. Primary study aims will yield proof-of-concept data on MIP feasibility and fidelity in usual care and evidence of MIP impact on psychiatric and behavioral services utilization, medication acceptance and compliance, and satisfaction with treatment services. Exploratory analyses will generate effect sizes for the short-term impact of MIP on the main targets of ADHD medication: ADHD symptoms and executive cognitive functioning. New study products would include a standardized and piloted MIP protocol, clinician training and fidelity monitoring procedures, and an observational fidelity instrument. If validated, MIP could be utilized as a stand-alone intervention in everyday care, or, be combined with existing manualized treatments for ASU in an effort to develop fully integrated treatment models for ASU/ADHD. Also, MIP could be delivered in conjunction with either family-based treatments or individual treatments that can flexibly include caregivers in early sessions.

ELIGIBILITY:
Inclusion Criteria:

* age 13-17, (2) caregiver able to participate in treatment,
* one day of alcohol use to intoxication or illegal drug use in the past 30 days (or 30 days prior to living in a controlled environment),
* endorsement of one or more DSM-IV symptoms of Substance Use or Alcohol Dependence/Abuse,
* meet ASAM criteria for outpatient substance use treatment,
* meet DSM-IV criteria for ADHD (with or without onset prior to age 7),
* not enrolled in any behavioral treatment.

Exclusion Criteria:

* MDD
* Bipolar Disorder
* mental retardation
* PDD
* medical or psychiatric illness requiring hospitalization
* current psychotic features
* current suicidality

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 14 (Actual)
Dates: Start 2011-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Medication Integration Protocol Feasibility, as assessed by qualitative interviewing of psychiatrist and therapists and also though qualitative interviews administered to teen and caregiver participants | Ongoing; 3-month follow-up
  Brief qualitative interviews will be designed and administered to the on-site psychiatrist and family therapists to capture judgments about the viability and acceptability of MIP compared to previous site practices, as well as its perceived short- and long-term safety and effectiveness for ASU/ADHD cases. A parallel qualitative interview will be administered to teens and caregivers at 3-month follow-up. MIP teens will also receive incentives to maintain medication diaries of daily pill intake, using the NIDA CTN method.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron T Hogue, PhD, Principal Investigator — The Natl Cntr on Addiction and Substance Abuse at Columbia University
Locations (1):
- Roberto Clemente Center, New York, New York, United States